CLINICAL TRIAL: NCT02196857
Title: Phase II Study of Sorafenib Plus 5-Azacitidine for the Initial Therapy of Patients With Acute Myeloid Leukemia and High Risk Myelodysplastic Syndrome With FLT3-ITD Mutation
Brief Title: Sorafenib Plus 5-Azacitidine Initial Therapy of Patients With Acute Myeloid Leukemia (AML) and High Risk Myelodysplastic Syndrome (MS) With FLT3-ITD Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0076; NCI-2014-01702 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Leukemia
Keywords: Leukemia; Acute myeloid leukemia; AML; High risk myelodysplastic syndrome; MDS; FLT3-ITD mutation; Azacytidine; 5-Azacytidine; 5-AZA; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Sorafenib; Nexavar; BAY 43-9006
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Azacitidine; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azacytidine + Sorafenib (Experimental): Azacitidine 75 mg/m2 administered subcutaneously (SQ) or intravenously (IV) daily for 7 days per 28 day cycle. Sorafenib administered orally at a dose of 400 mg twice daily every day continuously.
  Interventions: Drug: Azacytidine; Drug: Sorafenib

INTERVENTIONS:
Drug: Azacytidine — 75 mg/m2 administered subcutaneously (SQ) or intravenously (IV) on Days 1 - 7 for a 28 day cycle.
  Other Names: 5-Azacytidine; 5-AZA; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
Drug: Sorafenib — 400 mg by mouth twice daily about 12 hours apart, every day for a 28 day cycle.
  Other Names: Nexavar; BAY 43-9006

SUMMARY:
The goal of this clinical research study is to learn if 5-azacitidine and sorafenib can help to control the disease in patients with Acute Myeloid Leukemia (AML) and high risk Myelodisplastic Syndrome (MDS) with FLT3-ITD mutation. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive 5-azacitidine either as an injection under the skin or by vein on Days 1-7 of each 28-day cycle. If by vein, the infusion will take about 10-40 minutes.

You will take sorafenib by mouth 2 times a day about 12 hours apart, with at least 1 cup (8 ounces) of water on an empty stomach, every day. If you vomit a dose, do not make it up. You should wait and take your next scheduled dose.

Each study cycle may last a little longer than 28 days, depending on how you are doing.

Study Visits:

Each week, blood (about 1 tablespoon) will be drawn for routine tests.

Each week for the first 6 weeks, and then as often as your doctor thinks it is needed, you will have your blood pressure measured.

Before each cycle, you will have a physical exam.

Before every 2-4 cycles, you will have a bone marrow aspirate to check the status of the disease.

Length of Study:

You may continue taking the study drugs for as long as your doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse or intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

End-of-Study Visit:

After you have stopped taking the study drugs, the following tests and procedures will be performed:

* You will have a physical exam.
* You will have a bone marrow aspirate to check the status of disease.
* Blood (about 2 tablespoons) will be drawn for routine tests.

Follow-Up Visits:

After your end-of-study visit, you will return to the clinic every 3 months and have the following tests and procedures:

* You will have a physical exam.
* Blood (about 2 tablespoons) will be drawn for routine tests.

This is an investigational study. Sorafenib is FDA approved and commercially available for the treatment of kidney cancer and liver cancer. 5-azacitidine is FDA approved for the treatment of MDS, but combining it with sorafenib is investigational. The study doctor can tell you how the study drugs are designed to work.

Up to 52 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with untreated AML (> or equal to 20% blasts in bone marrow and/or peripheral blood) or high risk MDS (> or equal to 10% blasts in bone marrow). A. Patients with AML and history of MDS who have received prior therapy with a hypomethylating agent (including azacytidine) and/or with lenalidomide for prior MDS are eligible if the treating physician feels that participation in the study is in the patients' best interest. B. Patients should have molecular evidence of the presence of FLT3-ITD mutation with a molecular burden of at least 10%.
2. Age > or equal to 60 years; patients younger than 60 who are unsuitable for or unwilling to receive standard cytotoxic chemotherapy are also eligible to be enrolled.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status < or equal 2.
4. Adequate liver (bilirubin < or equal to 1.5 x ULN, Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) < or equal to 2.5 x ULN and Alkaline phosphatase < or equal to 4 x ULN if not related to leukemic disease) and renal (creatinine < or equal to 1.5 x ULN) function.
5. Patients must provide written informed consent.
6. Patients must have been off therapy for MDS for 2 weeks prior to entering this study, and must have recovered from the toxic effects of that therapy to at least grade 1, unless there is evidence of rapidly progressive disease. Use of hydroxyurea (any dose) or ara-C (up to 1 g/m^2 X 2 doses) for patients with rapidly proliferative disease is allowed before the start of study therapy; these should be stopped for 24 hours prior to the initiation of azacitidine and sorafenib.
7. Women of childbearing potential should be advised to avoid becoming pregnant with an adequate method of contraception (barrier or hormonal methods) and men should be advised to not father a child while receiving treatment with azacitidine. All men and women of childbearing potential must use acceptable methods of birth control throughout the study as described below: Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment. Men should use adequate birth control for at least 30 days after the last administration of sorafenib. Post-menopausal women (defined as no menses for at least one year) and surgically sterilized women are not required to undergo a pregnancy test. Females of childbearing potential: Recommendation is for 2 effective contraceptive methods during the study.
8. 7. Continued: Adequate forms of contraception are double-barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral, depo provera, or injectable contraceptives, intrauterine devices, and tubal ligation. Male patients with female partners who are of childbearing potential: Recommendation is for male and partner to use at least 2 effective contraceptive methods, as described above, during the study.
9. Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
10. International Normalized Ratio (INR) < or equal to 1.5. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored weekly, or as defined by the local standard of care, until INR is stable.

Exclusion Criteria:

1. Nursing and pregnant females.
2. Patients with acute promyelocytic leukemia are excluded.
3. Patients with known allergy to sorafenib or azacitidine, mannitol or any of their components.
4. Patients with known severe impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of sorafenib.
5. Patients with any other known disease (except carcinoma in-situ) or concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, cardiovascular disease including congestive heart failure, myocardial infarction within 6 months and uncontrolled hypertension, chronic renal disease (creatinine clearance < 20 ml/min using the Cockcroft and Gault formula), or active uncontrolled infection) which could compromise participation in the study.
6. Patients with a known confirmed diagnosis of HIV infection or active viral hepatitis (B or C).
7. Patients who have had any major surgical procedure within 28 days prior to Day 1.
8. Patients unwilling or unable to comply with the protocol.
9. Cardiac disease: Congestive heart failure > class II New York Heart Association (NYHA). Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
10. Uncontrolled hypertension defined as systolic blood pressure > 150? mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
11. Active clinically serious infection > CTCAE v4, Grade 2 not controlled with antibiotics.
12. Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
13. Pulmonary hemorrhage/bleeding event > or equal to CTCAE v4. Grade 2 within 4 weeks of first dose of study drug.
14. Any other hemorrhage/bleeding event > or equal to CTCAE v4. Grade 3 within 4 weeks of first dose of study drug.
15. Serious non-healing wound, ulcer, or bone fracture.
16. Evidence of bleeding diathesis or coagulopathy within the past 6 months.
17. Known or suspected allergy to sorafenib or any agent given in the course of this trial.
18. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results including known non-compliance issues on study trials.
19. Use of strong CYP3A4 inducer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02-06 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ohanian M, Garcia-Manero G, Levis M, Jabbour E, Daver N, Borthakur G, Kadia T, Pierce S, Burger J, Richie MA, Patel K, Andreeff M, Estrov Z, Cortes J, Kantarjian H, Ravandi F. Sorafenib Combined with 5-azacytidine in Older Patients with Untreated FLT3-ITD Mutated Acute Myeloid Leukemia. Am J Hematol. 2018 Sep;93(9):1136-1141. doi: 10.1002/ajh.25198. Epub 2018 Aug 31. PMID 30028037
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 2015 - February 2018
Period: Overall Study
Arm/Group | Azacytidine + Sorafenib
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Azacytidine + Sorafenib
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 16
Age, Continuous [Median (Full Range); unit: years] | 75 [67 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Response CR + PR + CRi
Description: Criteria for response per the International Working Group for myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML). Complete Response (CR) was defined as </= 5% blasts in the bone marrow (BM) with peripheral blood (PB) demonstrating greater thatn 1x10^9/L platelets with no detectable extramedullary disease. CR with incomplete recovery of PB counts (CRi) is the above criteria but neutrophil or platelet counts less than the stated values. Partial Response (PR) required all of the hematologic values for a CR but with a reduction of at least 50% in the percentage of blasts to 5% to 25% in the bone marrow aspirate.
Time Frame: After 3, 28 day cycles
Measure: Count of Participants; unit: Participants
Arm/Group | Azacytidine + Sorafenib
Number analyzed (Participants) | 16
Participants
  Complete Response (CR) | 4
  Partial Response (PR) | 1
  CR with incomplete platelet recovery (CRi) | 4

2. Secondary Outcome: Toxicity Profile of Azacytidine and Sorafenib
Description: Severity of toxicities graded according to the NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0. Standard reporting guidelines followed for adverse events. Safety data summarized by category, severity and frequency.
Time Frame: After 3, 28 day cycles
Measure: Count of Participants; unit: Participants
Arm/Group | Azacytidine + Sorafenib
Number analyzed (Participants) | 6
Participants
  Diarrhea | 4
  Dyspnea | 2
  Fatigue | 5
  Febrile Neutropenia | 4
  Nausea | 2
  Pain | 2
  Rash/Desquamation | 2

ADVERSE EVENTS:
Time Frame: Up to three years
Arm/Group | Azacytidine + Sorafenib
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 14/16
Other Adverse Events (participants affected / at risk) | 6/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacytidine + Sorafenib (N=16)
Acute Heart Failure (Cardiac disorders) | 1 (1)
Acute Kidney failure (Renal and urinary disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac Triponin Increase (Blood and lymphatic system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2)
Colitis (Gastrointestinal disorders) | 2 (4)
Dehydration (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Facial Pain/Dental (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Febrile Neutropenia (Infections and infestations) | 5 (8)
Fever (General disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Hypotnesion (Vascular disorders) | 4 (4)
Infection (Infections and infestations) | 1 (1)
Intestine Obstruction (Gastrointestinal disorders) | 1 (1)
Intracranial Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Laryngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Lung Infection (Infections and infestations) | 5 (12)
generalized edema (Renal and urinary disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacytidine + Sorafenib (N=16)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1)
Dyspena (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (5)
Hemorrhage (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Watery eye (Eye disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT02196857/Prot_SAP_000.pdf